CLINICAL TRIAL: NCT05838482
Title: Clinical Feasibility and Evaluation of Silicon Photon Counting CT
Status: Recruiting | Type: Observational
Sponsor: GE Healthcare (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 23000861577
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: CT Photon-Counting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subject's Scanned with Investigational Device: Eligible and consented subjects will be scanned using the investigational Pluto Photon-Counting CT system.
  Interventions: Device: CT Photon-Counting

INTERVENTIONS:
Device: CT Photon-Counting — Enrolled subjects will complete an exam using the photon-counting CT, with or without IV contract as indicated. Images will then be compared with the previously acquired CT conducted as standard of care.

SUMMARY:
The purpose of the study is to collect data to evaluate utility of the using photon-counting CT in a clinical setting.

DETAILED DESCRIPTION:
Data collected in this study includes an assessment of image quality parameters including spatial resolution, image contrast, and noise that will evaluate the product and how this photon-counting CT technology can be used to reduce the overall radiation dose in CT imaging, and enhance clinical applications for CT technology. This data and analysis will help support regulatory submission.

ELIGIBILITY:
Inclusion Criteria:

* Who are 18 years of age or older
* Able to sign and date the informed consent form
* Who have in the past 120 days or will in the future 30 days undergo a clinically-indicated CT exam of the head, neck, heart, chest, abdomen, pelvis, or extremities where images are available for this prior scheduled exam

Exclusion Criteria:

* Who are pregnant or lactating;
* Who were previously enrolled in this study;
* For contrast-enhanced CT exams, anyone with known or suspected allergy to iodinated contrast agents
* For contrast-enhanced CT exams, anyone with known or suspected renal insufficiency as determined by site medical personnel;
* Who need urgent or emergent care;
* Who have any conditions that, in the opinion of the PI or designee, would interfere with the evaluation of the results or constitute a health hazard for the subject; OR
* Who are unwilling to have GEHC personnel present for the CT exam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subject population will consist of adults that are 18-years of age or older, and who have undergone a prior clinically-indicated CT exam of at least one of the following anatomical area(s): head, neck, heart, chest, abdomen, pelvis, and/or extremities.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Data Collection | 1 year
  Number of Participants with raw investigational photon-counting CT scan data along with prior standard of care diagnostic CT exam data/images

SECONDARY OUTCOMES:
Image Quality | 1 year
  Reconstructed images produced from the raw investigational photon-counting CT scan will be scored for image quality using a Likert Scale (1 - Non-Diagnostic to 5 - Excellent Image Quality)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Thomsen, Study Director — GE Healthcare
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Scan data will be shared with other researchers but all will be completely deidentified.